CLINICAL TRIAL: NCT03165890
Title: Effect of Acetazolamide on Visuomotor Learning Performance in Patients With Chronic Obstructive Pulmonary Disease at Altitude
Brief Title: Effect of Acetazolamide on Cognition in Patients With Respiratory Disease at Altitude
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: National Center of Cardiology and Internal Medicine named after academician M.Mirrakhimov (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2017-00137A
Record Dates: First submitted 2017-05-23; First posted 2017-05-24 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: cognition; visuomotor learning; airway disease; altitude; prevention; acetazolamide
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Acetazolamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACETAZOLAMIDE oral capsule (Active Comparator): Acetazolamide 375mg/day (capsule @125 mg: 1 in the morning, 2 in the evening), orally. Medication starts 24 hours before ascent to 3200m until the morning after the second night at 3200m
  Interventions: Drug: ACETAZOLAMIDE oral capsule
- PLACEBO oral capsule (Placebo Comparator): Placebo (capsules identically looking as acetazolamide capsules: 1 in the morning, 2 in the evening), orally. Medication starts 24 hours before ascent to 3200m until the morning after the second night at 3200m.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: ACETAZOLAMIDE oral capsule — Administration of 125mg acetazolamide in the morning, 250mg in the evening, starting 24 hours before departure to 3200m
  Arms: ACETAZOLAMIDE oral capsule
Drug: Placebo oral capsule — Administration of equally looking placebo capsules in the morning and evening, starting 24 hours before departure to 3200m
  Arms: PLACEBO oral capsule

SUMMARY:
Randomized, placebo controlled trial evaluating the effect of acetazolamide on cognition in lowlanders with chronic obstructive pulmonary disease travelling from 760 m to 3200 m.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blind parallel trial evaluating the effect of acetazolamide (375 mg per day) vs. placebo on visuomotor learning performance at altitude (Tuja Ashu, 3200 m). Randomization to acetazolamide or placebo will be carried out after baseline measurements in Bishkek (760 m).

Visuomotor learning performance will be tested by Motor Task Manager (MTM). The MTM requires the subjects to reach visual targets with a hand-held cursor. During progression of the test, the movement direction from the cursor on the computer screen will increasingly differ from the direction of the hand movement, forcing the unaware subject to implicitly adapt to the imposed cursor rotation. This test assesses a subjects ability to visuomotor adaption, perception and attention. Furthermore, as the task will be performed in the evening and after sleep in the next morning, the investigators will be able to assess overnight improvement of implicit learned skills.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, age 18-75 yrs.
* COPD diagnosed according to GOLD, FEV1 40-80% predicted, SpO2 ≥92% at 750 m.
* Born, raised and currently living at low altitude (<800m).
* Written informed consent.

Exclusion Criteria:

* COPD exacerbation, very severe COPD with hypoxemia at low altitude (FEV1/FVC <0.7, FEV1 <40% predicted, oxygen saturation on room air <92% at 750 m).
* Comorbidities such as uncontrolled cardiovascular disease, i.e., unstable systemic arterial hypertension, coronary artery disease; previous stroke; OSA; pneumothorax in the last 2 months.
* Internal, neurologic, rheumatologic or psychiatric disease including current heavy smoking (>20 cigarettes per day)
* Known renal failure or allergy to acetazolamide and other sulfonamides

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2017-07-24 (Actual); Study Completion 2017-07-24 (Actual)

PRIMARY OUTCOMES:
visuomotor learning performance, drug effect | Day 2 at 760m and 3200m
  Difference in altitude-induced change in directional error between acetazolamide and placebo group, measured by the motor task manager
visuomotor learning performance, altitude effect | Day 1 and 2 at 760 m and at 3200m
  Difference in directional error between 760 m and 3200 m altitude in placebo group

SECONDARY OUTCOMES:
arterial oxygen saturation | Day 1 and 2 at 760 m and at 3200m
  Difference in altitude-induced change of arterial oxygen saturation between acetazolamide and placebo group, measured by pulse oxymetry

CONTACTS AND LOCATIONS:
Overall Officials: Konrad E Bloch, MD, Study Chair — University of Zurich; Talant M Sooronbaev, MD, Study Director — National Center of Cardiology and Internal Medicine, Bishkek, Kyrgyzstan
Locations (1):
- National Center of Cardiology and Internal Medicine, Bishkek, Kyrgyzstan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Scheiwiller PM, Furian M, Buergin A, Mayer LC, Schneider SR, Mademilov M, Lichtblau M, Muralt L, Sheraliev U, Sooronbaev TM, Ulrich S, Bloch KE. Visuomotor performance at high altitude in COPD patients. Randomized placebo-controlled trial of acetazolamide. Front Physiol. 2022 Sep 8;13:980755. doi: 10.3389/fphys.2022.980755. eCollection 2022. PMID 36160864